CLINICAL TRIAL: NCT06475677
Title: Prospective Trial of the OrthoCor Advanced System for Patients With Knee Osteoarthritis
Brief Title: OrthoCor Advanced Trial for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Caerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REP-152
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis, Knee; Osteo Arthritis Knee
Keywords: PEMF; Pulsed ElectroMagnetic Field
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: As osteoarthritis is a chronic condition, outcomes will be compared to baseline measurements for the same participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- OrthoCor Advanced System (Experimental): The OrthoCor Advanced System's novel combination of PEMF with the ability to monitor mobility metrics may have additional beneficial effects on pain, function, and quality of life for individuals affected by osteoarthritis.
  Interventions: Device: OrthoCor Advanced System

INTERVENTIONS:
Device: OrthoCor Advanced System — The OrthoCor Advanced System is a portable battery-operated non-invasive device that delivers Pulsed Electromagnetic Field (PEMF) plus heat therapy for general use pain relief. It utilizes a wrap that positions the device over painful areas and joint motion tracking recorded by a smart device application to monitor recovery metrics and therapy compliance.

SUMMARY:
The objective of this clinical trial is to show that PEMF therapy, heat, recovery metrics, and compliance data provided by the OrthoCor Advanced System improves pain and quality of life for patients with osteoarthritis. The main question it aims to answer is:

Does therapy from the OrthoCor Advanced System improve symptoms of osteoarthritis?

Researchers will compare range of motion measurements, sit to stand test results, and functional survey answers to see if there are any changes after 4 weeks of therapy with the OrthoCor Advanced System.

Participants will use the OrthoCor Active System for 30 minutes twice daily and complete recovery measurements daily using an application.

DETAILED DESCRIPTION:
Osteoarthritis is a chronic condition characterized by degeneration of the joints, affecting up to 240 million people worldwide.1 Its disabling effects are frequently associated with persistent joint pain, loss of mobility and function, and decreased quality of life that often lead to surgical procedures such as partial or total joint arthroplasty.1 Pulsed Electromagnetic Field (PEMF) therapy is a safe, clinically proven, nonpharmacological therapy that has previously been shown to have beneficial effects on pain and physical function in patients with osteoarthritis.1,2 The OrthoCor Advanced System's novel combination of PEMF with the ability to monitor mobility metrics may have additional beneficial effects on pain, function, and quality of life for individuals affected by osteoarthritis.

PEMF is a low-level, time-varying electromagnetic field that passes through and affects superficial soft tissue, helping to accelerate the body's natural anti-inflammatory and recovery responses. PEMF has been shown to stimulate tissue repair pathways that result in pain and inflammation reduction, such as the binding of calcium (Ca2+) to calmodulin (CaM) which triggers an anti-inflammatory nitric oxide (NO) cascade.2-4 NO is a key element in the body's natural healing process. It is also a vasodilator, increasing blood and lymphatic flow.3 Additionally, NO down-regulates interleukin-1 beta (IL1β) and inducible nitric oxide synthase (iNOS), which leads to reduced cyclooxygenase-2 (COX-2) activation and fewer prostaglandins - molecules responsible for causing inflammation and pain.5 Unlike other systemic COX-2 inhibitors such as nonsteroidal anti-inflammatory drugs (NSAIDs), OrthoCor's targeted PEMF signals locally modify these pathways, thereby reducing pain and inflammation without the risks and side effects associated with systemic medication.5

In addition to applying PEMF therapy, the OrthoCor Advanced System features a consumer facing smart device application as well as prescriber portal, allowing direct visibility of therapy compliance, reported pain levels, and functional performance metrics by both patient and physician. Daily recovery measurements may additionally supplement range of motion and joint strengthening and may encourage daily adherence to prescribed physical therapy and exercise. Strengthening exercises are considered a core standard of care treatment for managing knee osteoarthritis.5 Thus, the combined effects of PEMF and recovery insights may provide enhanced benefits to affected patients.

The OrthoCor Advanced System is a portable (battery operated) non-invasive device that delivers Pulsed Electromagnetic Field (PEMF) therapy plus chemical heat from OrthoPods for pain relief in the ankle, back, knee, wrist, elbow, shoulder, foot, or neck, while also providing the user with functional and mobility metrics. The microprocessor delivers the pulsed RF signal to the tissue target via inductive coupling with an applicator coil, while a 9-axis motion sensor tracks joint mobility during therapy.

The objective of this study is to evaluate the effectiveness of the OrthoCor Advanced System device for relieving symptoms and improving physical function in patients with osteoarthritis of the knee. It is hypothesized that the OrthoCor Advanced System device will improve knee range of motion and reported quality of life, as well as decrease reported pain levels associated with the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting to the study site with knee pain for at least 3 months, with articular cartilage loss confirmed by imaging study
2. An initial pain VAS score >4
3. At least 2 hours of daily standing and/or walking activity
4. Prescribed use of the OrthoCor Advanced System
5. Daily access to a smartphone or tablet compatible with the OrthoCor Medical application
6. Able to download and install app to smart phone
7. Willing and able to provide written consent
8. ≥18 years of age

Exclusion Criteria:

1. Previous diagnosis of rheumatoid arthritis or gout
2. Cortisone injection, knee surgery, or viscosupplementation in the previous 6 months
3. Prior knee replacement
4. Have a cardiac pacemaker, cardioverter defibrillator, neurostimulator, infusion pump or any active medical implant
5. Have an implanted metallic lead or any type of wire coil implant, or any implanted system that may contain a lead
6. Known or expected pregnancy
7. Have an open wound at the area of application
8. Are not able to sense or not fully aware of the sensation of heat
9. Have poor circulation or heart disease
10. Have uncontrolled diabetes
11. Under the age of 18 or individuals with open bone growth plates
12. Unwilling or unable to provide written consent
13. Unwilling or unable to use the OrthoCor Advanced System
14. Unwilling or unable to complete the pain assessment survey
15. Enrolled in a study to evaluate an investigational drug
16. Prisoner or under incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events | during 4 weeks of treatment
  Primary Safety Endpoint: Number of Adverse Events
VAS pain score | before, during, and after 4 weeks of treatment
  Primary Efficacy Endpoint: Pain score from 0-10 on the Visual Analog pain Scale (VAS), with 0 indicating no pain and 10 indicating the worst pain imaginable

SECONDARY OUTCOMES:
Knee AROM | before and after 4 weeks of treatment
  Active Range of Motion (AROM) for the Knee
Sit-to-stand | before and after 4 weeks of treatment
  Number of times in 30 seconds patient can perform sit-to-stand motion
KOOS survey | before and after 4 weeks of treatment
  Knee injury and Osteoarthritis Outcome Score (KOOS) survey, from 0-100% with 0% indicating the worst function possible and 100% indicating full function
Pain medication use | during 4 weeks of treatment
  Daily recording of pain medication taken
Joint motion tracking | during 4 weeks of treatment
  Joint motion tracking data recorded by the application during daily recovery exercises

CONTACTS AND LOCATIONS:
Overall Officials: Joshua G Hackel, MD, Principal Investigator — The Andrews Research & Education Foundation
Locations (1):
- Andrews Research & Education Foundation, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No